CLINICAL TRIAL: NCT04103151
Title: Rapid Triage for Serious Infections in Infants Younger Than 3 Months Using A Novel Heart Rate Variability Tool
Brief Title: Heart Rate Variability in Febrile Young Infants
Acronym: HRV
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: HRV-INFANTS-2017
Record Dates: First submitted 2019-09-08; First posted 2019-09-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Heart Rate; Variability; Triage; Decision Support Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Febrile infants: Febrile Infants less than 3 months presenting to the emergency department with a temperature of ≥ 38oC.
  Interventions: Device: Single lead ECG
- Afebrile infants: Afebrile Infants less than 3 months presenting to the emergency department
  Interventions: Device: Single lead ECG

INTERVENTIONS:
Device: Single lead ECG — Heart Rate Variability will be monitored using a single lead electrocardiogram

SUMMARY:
Febrile infants younger than 3 months old present a diagnostic dilemma to the emergency physician. Tension remains between the need for early aggressive intervention among patients with suspected sepsis and the global phenomena of increasing antibiotic resistance.

The investigators aim to: (1) To study the association between heart rate variability (HRV) and the presence of a serious infection (SI) among infants younger than 3 months old. The investigators hypothesize that a reduced HRV is associated with the presence of SI. (2) To compare HRV between febrile infants < 3 months with non-febrile infants. The investigators hypothesize that the variability will be reduced in febrile infants with SIs when compared to non-febrile well infants, but not among febrile infants without SIs when compared to non-febrile well infants. (3) To study if HRV will provide incremental diagnostic information over current triage tools.

DETAILED DESCRIPTION:
Febrile young infants younger than 3 months old present a diagnostic dilemma to the pediatric emergency department (ED) physician. The potential for a missed serious infection (SI) poses the threat of premature death and long-term disability among these infants. Despite decreasing early-onset neonatal sepsis rates due to obstetric prevention strategies, high rates of hospitalization and administration of parenteral antibiotics occur in this age group. Continual tension remains between the need for early and aggressive intervention among patients suspected with sepsis and the global phenomena of increasing antibiotic resistance. Research networks have attempted to build diagnostic algorithms to guide the identification of these ill infants. These are often useful as adjuncts to the clinician's gestalt, but generalizability remains questionable.

Vital signs are of paramount importance in recognizing ill children and have been used in pediatric early warning system scores (PEWS) and various triage systems. Vital signs have resurfaced as the focus of research in recent years, with various groups purposing to update evidence-based normal heart rate ranges among children. Normative heart rate ranges are infamously difficult to define due to the hemodynamic lability in these young infants, multiple confounders for abnormal heart rate, and the variable physiological response during acute stress states.

Previous pilot data showed that the Advanced Paediatric Life Support (APLS) and Fleming (<10th or >90th centile) guidelines performed with the highest sensitivity (66.0% and 62.6%, respectively) and the highest Negative Predictive Value (NPV) (73.3% and 71.4%, respectively). No single guideline reached a sensitivity of greater than 70%.

Objectives and Hypothesis

1. To study the association between heart rate variability (HRV) and the presence of a serious infection (SI) among infants younger than 3 months old. The investigators hypothesize that a reduced HRV is associated with the presence of SI.
2. To compare HRV between febrile infants < 3 months with non-febrile infants. The investigators hypothesize that the variability will be reduced in febrile infants with SIs when compared to non-febrile well infants, but not among febrile infants without SIs when compared to non-febrile well infants.
3. To study if HRV will provide incremental diagnostic information over current triage tools.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 3 months presenting to the ED will be included (both febrile and non-febrile) Febrile infants are those with an axillary or rectal temperature ≥ 38oC at triage and/or outside of the hospital. OR Non-febrile infants include those presenting to the ED for serum bilirubin checks or otherwise

Exclusion Criteria:

* Infants who are in active resuscitation for septic shock. Infants of parents who refused to give informed consent. Premature infants delivered at a gestation of < 35 weeks.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 330 infants < 3 months presenting with fever. Fever is defined as an axillary or rectal temperature ≥ 38oC.
  75 infants < 3 months (clinically well) presenting without fever. These include young infants presenting for neonatal jaundice or other non-febrile conditions.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with Serious Infections | Within 2 weeks of hospitalisation
  Serious infections are defined by: Sepsis, meningitis, lobar pneumonia, osteomyelitis, abscess, and urinary tract infection

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children' Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared with current study team. Sharing of de-identified data with collaborators will be reviewed by the study team.

REFERENCES:
- [Derived] Choa ZX, Raveentheran G, Khoo ZX, Ong GY, Wong L, Piragasam R, Ganapathy S, Chong SL. Prevalence of serious bacterial infections and performance of inflammatory markers in febrile infants with and without proven viral illness. Emerg Med J. 2025 Oct 20;42(11):721-727. doi: 10.1136/emermed-2024-214435. PMID 40335269
- [Derived] Chong SL, Ong GY, Allen JC, Lee JH, Piragasam R, Koh GZX, Mahajan P, Liu N, Ong MEH. Early prediction of serious infections in febrile infants incorporating heart rate variability in an emergency department: a pilot study. Emerg Med J. 2021 Aug;38(8):607-612. doi: 10.1136/emermed-2020-210675. Epub 2021 Apr 16. PMID 33863774